CLINICAL TRIAL: NCT07131280
Title: National Collaborative Centre for Hepatic Regenerative Medicine(NC-CHRM): To Study the Efficacy of Single vs Repeated Cycle of GCSF+ Darbepoetin in Long Term Transplant Free Management of Patient With Early Decompensated Cirrhosis
Brief Title: National Collaborative Centre for Hepatic Regenerative Medicine (NC-CHRM): Single vs Repeated Cycle of Granulocyte Colony-Stimulating Factor (GCSF) & Darbepoetin in Early Decompensated Cirrhosis
Acronym: NC-CHRM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Collaborators: Indian Council of Medical Research (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-Cirrhosis-75
Record Dates: First submitted 2025-07-11; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Decompensated Cirrhosis
Keywords: GCSF; Decompensated cirrhosis; Darbepoetin
MeSH Terms: interventions — Granulocyte Colony-Stimulating Factor; Darbepoetin alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Three cycles of GCSF+ darbepoetin and standard medical treatment (Experimental): Patient randomize for Three cycle of GCSF+ darbepoetin together with standard medical treatment, G-CSF will be given at a dose of 5 μg/kg s/c at days 1, 2, 3, 4, 5 and then every third and 7th day till day 30 based on hematological response and darbepoetin will be given s/c at dose of 40mcg once a week (total 4 doses) for 1 month. Second cycle of GCSF+ darbepoetin will be given after 1 month of completion of first cycle that is at month 3 and third cycle will be given 1 month after completion of 2nd cycle that is at 5th month. All patients will receive the standard medical treatment.
  Interventions: Drug: Gcsf; Drug: Darbepoetin; Other: Standard Medical Treatment
- Single cycle of GCSF+ darbepoetin and standard medical treatment (Active Comparator): Patient randomize for Single cycle of GCSF+ darbepoetin together with standard medical treatment, G-CSF will be given at a dose of 5 μg/kg s/c at days 1, 2, 3, 4, 5 and then every third and 7th day till day 30 based on hematological response and darbepoetin will be given s/c at dose of 40mcg once a week (total 4 doses) for 1 month. All patients will receive the standard medical treatment.
  Interventions: Drug: Gcsf; Drug: Darbepoetin; Other: Standard Medical Treatment

INTERVENTIONS:
Drug: Gcsf — G-CSF will be given at a dose of 5 μg/kg s/c at days 1, 2, 3, 4, 5 and then every third and 7th day till day 30
Drug: Darbepoetin — Darbepoetin will be given s/c at dose of 40mcg once a week for 1 month
Other: Standard Medical Treatment — Standard Medical Treatment

SUMMARY:
Chronic liver disease is a growing health concern, with limited access to liver transplants. This study addresses the urgent need for alternatives by exploring regenerative therapies, like G-CSF, to boost the liver's natural repair. The goal is to develop safe, effective, and accessible treatments for patients who cannot undergo transplant.

DETAILED DESCRIPTION:
The incidence of deaths from chronic liver diseases (CLD) and cirrhosis are rapidly increasing globally, including India. Liver transplant is the only curative option. Unfortunately, transplant is often not feasible. There is a need for nearly 100,000 liver transplants every year in India, though, only about 2,500 transplants are being done at present across the country. There is therefore, a huge unmet need of developing non-transplant options for chronic liver disease patients. In this regard emerging science of regenerative therapy holds great promises but therapeutic benefit of these therapies is limited due to lack of clinical validation.

Novelty: Cirrhosis as a result of hepatitis B and C can regress with effective antiviral therapy. Therapeutic options for patients with cryptogenic or alcoholic cirrhosis are, however, limited. With limited options for transplant. Liver failure is failure of regeneration hence, potentiating native liver repair and regeneration can serve as potential non-transplant approaches. Growth factors {like GCSF, darbepoetin (EPO) have shown survival benefits with improve liver repair and regeneration in clinical trials by us (Gastroenterology 2012, 2015, Liver Int. 2019; Hepatology 2021) and others, however the effect is transient. In the proposed National Collaborative Centre for Hepatic Regenerative Medicine (NC-CHRM) we will use this novel regenerative medicine approaches GCSF therapy (for management of chronic liver failure) to develop safe and effective regenerative therapy clinical protocol for transplant free management of liver failure in cirrhosis. Using integrated cellular, molecular and functional analysis we will also establish their mechanism of action and identify biomarker to access therapeutic response.

ELIGIBILITY:
Inclusion Criteria:

* Early decompensated cirrhosis patients with MELD <16

Exclusion Criteria:

* Patients with age less than 18 years or more than 65 years
* Patients with Grade III ascites
* CHILD C cirrhosis
* Patients with a known focus of sepsis; spontaneous Bacterial Peritonitis (SBP)
* variceal bleeding in past 3months
* Hepatocellular Carcinoma (HCC) or other malignancy
* Acute Kidney Injury (AKI) with serum Creatinine >1.5 mg/ dl, multi-organ failure, grade 3 or 4 Hepatic Encephalopathy (HE),
* HIV seropositivity
* Medically uncontrolled essential hypertension
* Pregnancy
* Viral etiology of liver disease
* Co-existent Hepatitis B, Hepatitis C, HIV
* Chronic kidney disease
* Lack of informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2031-07 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Transplant-free survival of GCSF + darbepoetin in patients with early decompensated cirrhosis in both groups. | 3 year

SECONDARY OUTCOMES:
Transplant-free survival | 6-month, one year, 2 year and 3 year
Proportion of patient developed new-onset of Liver Related Event (such as ascites, hepatic encephalopathy , acute kidney injury, bleed and sepsis) or show mortality in both the groups | 6-month, one year, 2 year and 3 year
Cumulative incidence of sepsis, acute kidney injury or secondary organ dysfunction in both groups | 6-month, one year, 2 year and 3 year
Cumulative incidence of second decompensation | 6-month, one year, 2 year and 3 year
Improvement in liver disease severity indices, including the Child-Turcotte-Pugh (CTP) score (ΔCTP). | 6-month, one year, 2 year and 3 year
Improvement in liver disease severity indice like Model for End-Stage Liver Disease (MELD) score (ΔMELD). | 6-month, one year, 2 year and 3 year
Proportion of patients completing treatment without major adverse effects | 6-month, one year, 2 year and 3 year
  Adverse effects will be graded in accordance to CTCAE
Impact on liver injury (assessed by AST and ALT levels in blood). | 6-month, one year, 2 year and 3 year
Impact on fibrosis (evaluated using Masson's Trichome stain and the Enhanced Liver Fibrosis [ELF] score). | 6-month, one year, 2 year and 3 year
Impact on regeneration (measured by plasma Alpha-Fetoprotein levels). | 6-month, one year, 2 year and 3 year
Impact on bone marrow stem cell reserve (CD34⁺ cell count in peripheral blood) | One year, 2 year and 3 year

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Shiv Kumar Sarin, DM, Principal Investigator — Institute of Liver & Biliary Sciences
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided